CLINICAL TRIAL: NCT03178214
Title: A Single Centre, Open-label, Randomised, Single Dose, Three-period, Crossover Study to Evaluate the Bioavailability of Infacort Administered as Sprinkles With Soft Food and Yoghurt Compared With Direct Administration to the Back of the Tongue in Dexamethasone-suppressed Healthy Adult Male Subjects
Brief Title: Bioavailability of Infacort When Administered Onto Food Compared to Direct Oral Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: Simbec Research (Industry); EMAS Pharma (Industry); Voet Consulting (Industry); Brush Clinical Research Ltd. (Industry); Medical Matters International Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Infacort 006
Record Dates: First submitted 2017-05-27; First posted 2017-06-06 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Infacort - Yoghurt (Experimental): One single 5mg dose of Infacort will be sprinkled onto 5mL of yoghurt and swallowed within three minutes. This will be taken with 240mL of water.
  Interventions: Drug: Infacort
- Infacort - Soft Food (Experimental): One single 5mg dose of Infacort will be sprinkled onto 5mL of soft food (such as applesauce) and swallowed within three minutes. This will be taken with 240mL of water.
  Interventions: Drug: Infacort
- Infacort - Dry Granules (Active Comparator): One single 5mg dose of Infacort will be administered as dry granules to the back of the tongue and swallowed. This will be taken with 240mL of water.
  Interventions: Drug: Infacort

INTERVENTIONS:
Drug: Infacort — Immediate-release multiparticulate formulation of hydrocortisone.

SUMMARY:
This is a single centre, open-label, randomised, single dose, three-period, crossover study to evaluate the bioavailability of Infacort® administered as 'sprinkles' with soft food and yoghurt compared with direct administration to the back of the tongue in dexamethasone-suppressed healthy adult male subjects.

The study will comprise of a pre-study screen, followed by 3 treatment periods and a post-study follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between 18 and 45 years of age, inclusive (at screening).
2. A BMI of 18-30 kg/m2 (inclusive).
3. No clinically significant abnormal serum biochemistry, haematology or urine examination values as defined by the Investigator.
4. A negative urinary drugs of abuse screen. A positive alcohol test may be repeated at the discretion of the Investigator.
5. Negative HIV and Hepatitis B and C results.
6. No clinically significant abnormalities in 12-lead ECG as defined by the Investigator.
7. No clinically significant deviation outside the normal ranges for blood pressure and heart rate measurements as defined by the Investigator (please refer to appendix 1 for normal ranges).
8. Subjects (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) and sexual partners must use 2 effective contraception methods during the trial and for 3 months after the last dose, for example:

   * Oral contraceptive + condom
   * Intra-uterine device (IUD) + condom
   * Diaphragm with spermicide + condom
9. Subjects must be available to complete all three periods of the study and the follow-up visit.
10. Subjects must satisfy a medical examiner about their fitness to participate in the study.
11. Subjects must be able to read and understand the informed consent form and must provide written informed consent to participate in the study.

Exclusion Criteria:

1. A clinically significant history of gastrointestinal disorder likely to influence drug absorption.
2. Receipt of any medication other than paracetamol within the 14 days prior to dosing (including topical steroids, high dose vitamins, dietary supplements or herbal remedies).
3. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
4. Receipt of any vaccination within the previous one month.
5. Presence of infections (systemic fungal and viral infections, acute bacterial infections).
6. Current or previous history of tuberculosis.
7. A clinically significant history of previous allergy/sensitivity to hydrocortisone, dexamethasone and/or any of the ingredients contained within the yoghurt or soft food (this includes lactose intolerance).
8. Meeting any of the contraindications for dexamethasone, as detailed in the Summary of Product Characteristics (SmPC).
9. A clinically significant history of drug or alcohol abuse.
10. Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
11. Participation in a New Chemical Entity or marketed drug clinical study within the previous 3 months or, five half-lives of study drug, whichever is the longer period. (NB. the three month washout period between trials is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
12. Subjects who have consumed more than two units of alcohol per day within seven days prior to the first dose or have consumed any alcohol within the 48-hour period prior to the first dose.
13. Donation or receipt of equal to/more than 450 mL of blood within the previous three months.
14. Subjects who smoke (or ex-smokers who have smoked within six months prior to first dose. This includes e-cigarette and shisha users).
15. Subjects who work shifts (i.e. regularly alternate between days, afternoons and nights).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) (0-t) of Infacort administered with yoghurt and soft food compared to dry granules administered to the back of the tongue | 12 hours post-IMP administration
  The pharmacokinetic parameter AUC0-inf of Infacort® administered as sprinkles with yoghurt and soft food compared to Infacort® administered as dry granules to the back of the tongue.
Area under the curve (AUC) (0-infinity) of Infacort administered with yoghurt and soft food compared to dry granules administered to the back of the tongue | 12 hours post-IMP administration
  The pharmacokinetic parameter AUC0-inf of Infacort® administered as sprinkles with yoghurt and soft food compared to Infacort® administered as dry granules to the back of the tongue.
Cmax of Infacort administered with yoghurt and soft food compared to dry granules administered to the back of the tongue. | Up to 12 hours post-IMP adminstration
  The pharmacokinetic parameter Cmax of Infacort® administered as sprinkles with yoghurt and soft food compared to Infacort® administered as dry granules to the back of the tongue.

SECONDARY OUTCOMES:
Tmax of Infacort® administered as sprinkles with yoghurt and soft food compared to Infacort® administered as dry granules to the back of the tongue. | Up to 12 hours post-IMP administration
  Tmax of Infacort® administered as sprinkles with yoghurt and soft food compared to Infacort® administered as dry granules to the back of the tongue.

CONTACTS AND LOCATIONS:
Locations (1):
- Simbec Research Ltd., Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No